CLINICAL TRIAL: NCT07262437
Title: Targeting Immunosuppressive Treatment for Non-infectious Uveitis Using Aqueous Humor Cytokine Profiles
Acronym: PRIN_NIU
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Alessandro Invernizzi, Professor of Ophthalmology, University of Milan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRIN_NIU
Record Dates: First submitted 2025-08-26; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-08

CONDITIONS: Uveitis Posterior Non-Infectious; Inflammation Eye; Uveitis; Uveitis, Anterior
Keywords: non-infectious uveitis; cytokines; aqueous humor; inflammation
MeSH Terms: conditions — Endophthalmitis; Uveitis; Uveitis, Anterior; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients affected by non-infective uveitis (Experimental): Those patients will be recruited from the routine clinical practice. The treatment choice is not pre-planned but it will be based on the treating physician's clinical decision.
  Interventions: Procedure: to improve clinical practice in treatment of non-infective uveitis

INTERVENTIONS:
Procedure: to improve clinical practice in treatment of non-infective uveitis — to identify the potential correlation between cytokine profiles and systemic immunosuppressive drug.

SUMMARY:
This multicenter, prospective, interventional, non-pharmacological study aims to investigate whether the intraocular cytokine profile is associated with the therapeutic response to immunosuppressive drugs in patients with non-infectious uveitis (NIU). Approximately 220 patients with NIU in at least one eye, showing inadequate response to topical or systemic corticosteroids at baseline and presenting with signs of anterior segment inflammation, will be enrolled to enhance sensitivity to laboratory assays. Aqueous humor and blood samples will be collected at baseline. Cytokine concentrations of 14 different cytokines will be measured using multiplex immunoassay techniques. Participants will receive immunosuppressive treatment based on standard clinical practice.

DETAILED DESCRIPTION:
This project is coordinated by University of Milan/ ASST FBF Sacco Milan Italy. Site coordinator has a sub-Unit (AUSL Reggio Emilia Italy) which act both as recruiter and Lab analyst.

Site co-partner is: IRCCS San Raffaele, University Vita e Salute San Raffaele Milan Italy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-infectious uveitis in at least one eye with incomplete or not sustained response to topic or systemic steroids at the baseline visit
* Evidence of anterior chamber inflammation to optimize lab sensibility
* As per clinical practice eligibility to receive one of the following immunosuppressive treatment: mycophenolate mofetil (MMF), methotrexate (MTX), azatioprine (AZA), adalimumab (ADA)
* Ability to provide informed consent

Exclusion Criteria:

* Concomitant immunosuppressive treatment
* Presence of other systemic pathologies that do not allow immunosuppressive therapies
* Ocular media opacities that could interfere with a good quality of fundus exam and/or imaging of the eye
* Any ocular or systemic condition that could interfere with cytokine profile expressions
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Aqueous humor cytokine profile characterization in responders vs non-responders using multiplex immunoassay techniques. | Three months from baseline
  Distribution of responders and non responders to each study drug according to baseline cytokine profile in the aqueous humor.

SECONDARY OUTCOMES:
Correlation cytokine profiles and patients' clinical evaluation | Baseline vs three months
  Correlation between patients' demographics, uveitis type, uveitis etiology, and duration with the cytokine profiles in the aqueous humor.
Correlation between clinical ophthalmic features and cytokine profiles | baseline and three months
  Correlation between clinical ophthalmic features and cytokine profiles in the aqueous humor.
Correlation between cytokine levels in the aqueous humor and blood | Baseline
  Comparison between cytokine levels in the aqueous humor and those in the plasma to identify differential expression in the two compartments.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Invernizzi, MD, Principal Investigator — University of Milan
Locations (3):
- Italy (3):
  - IRCCS San Raffaele Università Vita e Salute, Milan
  - ASST Fatebenefratelli Sacco P.O.L.Sacco, Milan
  - AUSL Reggio Emilia, Reggio Emilia

IPD SHARING:
Plan to Share IPD: Yes
Each site will be co-owner of IPD. Date will be disclosed in aggregated form